## Appendix Z. Consent- Participant Satisfaction Interview

### RESEARCH INFORMED CONSENT

# One-on-One Interview with Research Participants in Group A – The Grow Well Program

**Study title:** GROW WELL/CRECER BIEN: Addressing Childhood Obesity in Low-income Families

**Investigator:** Ann Cheney, PhD, Associate Professor, Dept. of Social Medicine Population and Public Health, School of Medicine, UC Riverside <a href="mailto:ann.cheney@medsch.ucr.edu">ann.cheney@medsch.ucr.edu</a>, (501) 352-8526.

**Community Investigator**: Maria Pozar, Conchita Servicios de la Comunidad, <u>pozarconchita@gmail.com</u>; 760-863-9432.

You have been invited to take part in a research project. It is described below. The researcher will explain the project. Feel free to ask questions. If you decide to participate, you will be asked to provide consent to participate in this study. This form will be a record of your agreement to participate. You will be given a copy of this form to keep.

**Important information about this study.** Below is some important information to know about this study. This information will help you decide if you want to participate or not. Carefully consider this information. Please ask any questions about anything you do not understand before you decide to participate.

## Why are we doing this study?

The purpose of the study is to see how well education material about infant growth supports Latino families caring for infants. The Grow Well team collaborated with mothers and caregivers to develop material to encourage families to raise healthy children. This study will tell us how well our program works, and if parents and caregivers are satisfied with the materials and activities.

**Eligibility for participation:** Participants in Group A- Grow Well of the study can participate in this interview. Participants must have completed the full six months of the study to be eligible to participate. You must be aged 18 years or older, and speak English, Spanish, or Purépecha.

**Procedures:** Participation in this part of the study will involve a one-time, one-on-one interview with you. The interview will last 30-60 minutes and will be conducted via Zoom or phone. In the interview the research team will ask for your feedback on the Grow Well material and program activity. We will ask you to share your thoughts about the program and satisfaction with the program. Such as what you thought about the in-person visits, phone call check ins, and WhatsApp posts. If you consent to audio recording, the interview will be audio recorded and trascribed. Go Transcript, a professional transcription service, will transcribe the recording. Go Transcript will not disclose any of your information or identify you. Our team will remove any personal information.

**Compensation:** You will receive a \$25 gift card for participating in the interview, at the end of the interview. There will be no out-of-pocket costs associated with study participation.



**Risks:** The risks of participation are minimal. You may worry whether your answers to the study questions are correct. However, there are no right or wrong answers to the questions. You can choose not to answer specific questions or take a brief break from data collection, if needed. There is a risk of a breach of confidentiality. We minimize this risk by using encryption and storing all data on a secure server and/or in a locked cabinet in a secure office, accessible only to the research team.

**Benefits:** Participation may provide the benefits of: 1) knowledge about how infant care and feeding shape child growth and potential risk for early childhood obesity, 2) knowledge about community-engaged participatory research, and 3) satisfaction with programs developed by mothers and caregivers for Latino families.

**Alternatives:** Your alternative to participating in this interview is not to participate.

**Voluntary participation:** Your participation in this study is voluntary. You can decide to participate or not to participate. You can decide to withdraw from the study at any point without penalty. Your choice about whether to participate or not to participate will not affect your employment or relationships with the UCR School of Medicine. To withdraw from the study, you would simply need to notify a research team member by phone, email, or in person, and the research team will destroy any data you have provided.

What happens to information collected for the research?: Your information collected as part of this research will be analyzed and shared with the community. It will also inform next steps for a larger study. Per the National Institutes of Health Data Management and Sharing Policy, we will make available for future research without your consent the material you share with us. All identifiers will be removed from the information you share. Your name will not be disclosed or linked to the data. All data will be maintained on secure servers at the University of California Riverside School of Medicine. The research team will delete personally identifying information (your name and contact information) once data collection is complete. It will delete audio recordings once research results are reported.

Will information about me be kept private? We will do our best to make sure that the personal information gathered for this study is kept private. However, we cannot guarantee total privacy. If required by the law, your personal information may be disclosed. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used. Authorized representatives from the following organizations may review your research data for the purpose of monitoring or managing the conduct of this study: UCR's Institutional Review Board, representatives of the National Institutes of Health, or representatives of the University of California.

Whom can I talk to? If you have questions, concerns, or complaints, or think the research has hurt you, talk to the investigators, named above. If you have questions about your rights or complaints as a research subject, please contact the IRB Chairperson at (951) 827-4802 during business hours, or by email at irb@ucr.edu.

### Consent

| Below, pleas | se indicate your cons | sent to participate in this interview. |
|---|---|---|
| Yes | Yes, I consent to participate in this interview. | |
| | [If yes, read] | Yes, I consent to be audio recorded. |
| No | No, I do not consent to participate in this interview. | |



| Printed name: |
|---|
| Date: |
| Please indicate your preference for receiving the gift card for your participation: |
| I prefer to receive the gift card by: |
| email (e-gift card). My email address is: |
| regular mail. My mailing address is: |
| delivered to my home. My home address is: |

